CLINICAL TRIAL: NCT06869031
Title: Construction and Verification of Adaptive Intervention Model for Self-Management Behavior of Hypertensive Patients in Rural Areas：A Perspective of Doctor-Patient Interactions
Brief Title: Adaptive Intervention Model for Hypertension Self-Management in Rural Areas: A Doctor-Patient Interaction Approach
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yuju Wu (Other)
Responsible Party: Sponsor-Investigator, Yuju Wu, Associate Professor, Sichuan University
Organization: Sichuan University (Other)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: Gwll2024130
Record Dates: First submitted 2025-02-19; First posted 2025-03-11 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Hypertension Self-management; Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Standard Interactive Intervention with Continued Standard Intervention for Poor Self-Management (Experimental): This study consists of two stage. In the first stage, participants are randomly assigned to the standard interactive intervention group. After six months, those with poor self-management behavior are randomly assigned to either continue the standard interactive intervention or switch to the enhanced interactive intervention in the second stage. This arm consists of participants who were initially assigned to the standard interactive intervention for six months and were subsequently reassigned to continue the standard interactive intervention in the second stage.
  The intervention content is designed based on the Health Behavior Interaction Model, covering four aspects: health information (e.g., potential risks of poor self-management behavior), professional skills (e.g., blood pressure measurement), emotional support (e.g., understanding the experiences of hypertension patients), and decision-making participation. Conducted once a month.
  Interventions: Behavioral: Standard Interactive Intervention for Hypertension Management
- Standard Interactive Intervention Followed by Enhanced Intervention for Poor Self-Management (Experimental): In the first stage, participants are randomly assigned to the standard interactive intervention group. After six months, those with poor self-management behavior are randomly assigned to either continue the standard interactive intervention or switch to the enhanced interactive intervention in the second stage. This arm consists of participants who were initially assigned to the standard interactive intervention for six months and were subsequently reassigned to the enhanced interactive intervention in the second stage.
  The enhanced interactive intervention refers to the same intervention as the standard interactive group, with an increased frequency of interactions. Every two weeks, a brief interactive intervention is conducted via the intelligent outbound call system to remind patients to perform their self-management behaviors.
  Interventions: Behavioral: Standard Interactive Intervention for Hypertension Management
- Standard Interactive Intervention Followed by Regular Follow-Up Management (Experimental): First phase: Randomly assigned to the standard interactive intervention group (6 months). Second phase: Participants with improved self-management behavior are transitioned to regular follow-up management (6 months).
  Interventions: Behavioral: Standard Interactive Intervention for Hypertension Management
- Intensified Interactive Intervention Followed by Standard Interactive Intervention (Experimental): In the first stage, participants are randomly assigned to the intensified interactive intervention group. After six months, those with improved self-management behavior are randomly assigned to either continue with the standard interactive intervention or transition to routine follow-up management. This arm consists of participants who were initially assigned to the intensified interactive intervention for six months and were subsequently reassigned to the standard interactive intervention in the second stage.
  Interventions: Behavioral: Intensified Interactive Intervention for Hypertension Management
- Intensified Interactive Intervention Followed by Routine Follow-Up (Experimental): In the first stage, participants are randomly assigned to the intensified interactive intervention group. After six months, those with improved self-management behavior are randomly assigned to either continue with the standard interactive intervention or transition to routine follow-up management. This arm consists of participants who were initially assigned to the intensified interactive intervention for six months and were subsequently reassigned to the routine follow-up management in the second stage.
  Interventions: Behavioral: Intensified Interactive Intervention for Hypertension Management
- Intensified Interactive Intervention with Continued Intensification (Experimental): In the first stage, participants are randomly assigned to the intensified interactive intervention group for six months. In the second stage, those with poor self-management behavior at the end of the first stage will continue receiving the intensified interactive intervention for another six months.
  Interventions: Behavioral: Intensified Interactive Intervention for Hypertension Management

INTERVENTIONS:
Behavioral: Standard Interactive Intervention for Hypertension Management — The standard interactive intervention is a doctor-patient interaction intervention conducted by follow-up physicians using an intelligent outbound call system as part of follow-up management. It is implemented once a month and is designed based on the Health Behavior Interaction Model, covering four key aspects: health information (e.g., potential risks of poor self-management behavior), professional skills(e.g., blood pressure measurement, medication guidance), emotional support , and decision-making participation.
  Arms: Standard Interactive Intervention Followed by Enhanced Intervention for Poor Self-Management; Standard Interactive Intervention Followed by Regular Follow-Up Management; Standard Interactive Intervention with Continued Standard Intervention for Poor Self-Management
Behavioral: Intensified Interactive Intervention for Hypertension Management — The enhanced interactive intervention builds upon the standard interactive intervention by increasing the frequency of interactions. In addition to the monthly intervention, patients receive an additional brief interactive intervention every two weeks via the intelligent outbound call system, reminding them to adhere to self-management behaviors for hypertension control.
  Arms: Intensified Interactive Intervention Followed by Routine Follow-Up; Intensified Interactive Intervention Followed by Standard Interactive Intervention; Intensified Interactive Intervention with Continued Intensification

SUMMARY:
The aim of this project is to develop and validate an adaptive intervention model to improve self-management behavior in rural hypertensive patients. The primary question it seeks to answer is: Can a tailored, interaction-based intervention model, guided by key doctor-patient interaction elements, effectively enhance self-management behavior among rural hypertensive patients and improve long-term blood pressure control? Researchers will evaluate the impact of different intervention strategies on self-management behavior and identify the most effective combination to establish a sustainable intervention model for rural hypertension management.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed hypertension patients who are permanent residents in rural areas.
* No plans for long-term relocation within the next year.
* Willing to participate in this study.
* No cognitive impairment.
* No other diseases that significantly affect self-management behavior, such as malignant tumors.

Exclusion Criteria:

* Age over 80 years.
* Having conditions such as stroke, paralysis, or mental disorders that prevent the completion of self-management behaviors.
* Severe hearing impairment or speech disorders that prevent participation in interviews.
* Likely to relocate or be away from the local area for an extended period within one year.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Hypertension self-management behavior | From the start of the intervention to the 6-month and the end of the trial at 12 months.
  Hypertension self-management behavior includes six dimensions: medication management, condition monitoring, dietary management, exercise management, work and rest management, and emotional management. Each item is scored on a 1 to 5 scale, with a total score ranging from 33 to 165. A higher total score indicates a higher level of self-management in patients.
Blood pressure | From the start of the intervention to the 6-month and the end of the trial at 12 months.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Fourth Hospital and West China School of Public Health. Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No